CLINICAL TRIAL: NCT02476097
Title: Study of the Effect of PROGRESSive Withdrawal Esomeprazole of on Acid-related Symptoms, PROGRESS Study A Randomized, Placebo-controlled, Double Blinded Study
Brief Title: PROGRESSive Withdrawal Esomeprazole and Acid-related Symptoms
Acronym: PROGRESS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Victoria Rollason (Other)
Responsible Party: Sponsor-Investigator, Victoria Rollason, Dr, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-003
Record Dates: First submitted 2015-06-15; First posted 2015-06-19 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Stomach Diseases
Keywords: esomeprazole randomized study; proton pump inhibitor; gastric acid rebound; randomized study; esomeprazole
MeSH Terms: conditions — Stomach Diseases | interventions — Esomeprazole; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sudden discontinuation (Placebo Comparator): placebo for 7 days
  Interventions: Other: CYP2C19 phenotypical analysis; Drug: Placebo
- Progressive discontinuation (Active Comparator): Esomeprazole: Nexium® 20mg, Astra Zeneca , for 7 days
  Interventions: Drug: Esomeprazole: Nexium® 20mg, Astra Zeneca; Other: CYP2C19 phenotypical analysis

INTERVENTIONS:
Drug: Esomeprazole: Nexium® 20mg, Astra Zeneca — Comparison of the prevalence of clinical symptoms of acid rebound, between patients with progressive (esomeprazole ) or sudden (placebo) discontinuation of Proton pump inhibitors.
  Other Names: Nexium®
  Arms: Progressive discontinuation
Other: CYP2C19 phenotypical analysis — All patients included will undergo an assessment of the CYP2C19 activity by the administration of omeprazole 40mg and following measurement of omeprazole metabolic ratio respectively, once during the study.
  Other Names: omeprazole 40mg
Drug: Placebo — Comparison of the prevalence of clinical symptoms of acid rebound, between patients with progressive (esomeprazole ) or sudden (placebo) discontinuation of Proton pump inhibitors.
  Arms: Sudden discontinuation

SUMMARY:
Rebound acid hypersecretion (RAHS), defined as an increase in gastric acid secretion above pre-treatment levels after PPIs therapy is observed within two weeks after withdrawal of treatment and could theoretically lead to acid-related symptoms such as heartburn, acid regurgitation, or dyspepsia that might result in resumption of therapy. A plausible physiologic theory for the rebound phenomenon suggests that long-term, elevated gastric pH caused by blockage of the proton-pumps stimulates compensatory gastrin release. Interestingly, Reimer et al. demonstrated the occurrence of RAHS in healthy volunteers who had received eight weeks of esomperazole. The clinical symptoms occured in a different prevalence compared with placebo treated patients at ten weeks after withdrawal and until the end of the study (twelve weeks). Twenty to twenty-two percent of patients displayed symptoms ten or twelve weeks after having discontinued PPIs while they occured in 1.7-7% of placebo-treated patients. Efforts should be pursued to restrict PPI therapy use to patients likely to benefit from it.

In this context, we propose to investigate the benefit of a progressive decrease in doses of esomeprazole compared to a sudden discontinuation. This is a randomized, double-blind, placebo-controlled trial with 156 patients treated by esomeprazole 40mg since four weeks least, randomized to one week of placebo or one week of esomeprazole 20mg. We want to compare the prevalence of clinical gastrointestinal symptoms between patients with progressive discontinuation (one week of esomeprazole, 20mg, then discontinuation) or those with sudden discontinuation of esomeprazole 40mg.

ELIGIBILITY:
Inclusion Criteria:

* Treatment by esomeprazole 40mg since 4 weeks or more
* Esomeprazole withdrawal decided by the clinician
* Male and female aged 18-90 years
* Volunteers to participate to the study
* Must understand and read French language
* Must be able to give a written informed consent

Exclusion Criteria:

* Impairment of cognitive status
* Current indication to continue PPI treatment
* History of erosive and ulcerative esophagitis, Barrett esophagus, Zollinger-Ellison syndrome
* Short-term treatment of documented ulcer disease, as part of a combination regimen for Helicobacter pylori (HP) eradication
* Prevention of ulcers due to non-steroidal anti-inflammatory drugs.
* Hepatic impairment (TP<60%)
* Hypersensitivity to omeprazole (CYP2C19 activity) or esomeprazole
* Current pregnancy or current breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-06; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The proportions of patients answering "yes" to the clinical gastrointestinal symptoms questions were comparable at visit 1. | day 8
  The five-item PASS test is a valid tool for the evaluation of persistent acid-related symptoms in patients receiving PPI therapy. It demonstrates good content validity, test-retest reliability, responsiveness and construct validity in both English and French forms. The PASS test is a simple, clinically applicable tool for the identification of patients with persistent acid-related symptoms during therapy and the assessment of their responses to a change in therapy.
  The investigators will modifiy the first question for the study. While, it is usually asked: " Are you taking prescription medication for any of the following stomach problems/symptoms:… " ; in the study, the investigators will ask : " Do you have any of the following stomach problems/symptoms : … ".
  With any of the 7 symptoms, the patient will be considered as symptomatic.
The proportions of patients answering "yes" to the clinical gastrointestinal symptoms questions were comparable at visit 2. | day 15
  The five-item PASS test is a valid tool for the evaluation of persistent acid-related symptoms in patients receiving PPI therapy. It demonstrates good content validity, test-retest reliability, responsiveness and construct validity in both English and French forms. The PASS test is a simple, clinically applicable tool for the identification of patients with persistent acid-related symptoms during therapy and the assessment of their responses to a change in therapy.
  The investigators will modifiy the first question for the study. While, it is usually asked: " Are you taking prescription medication for any of the following stomach problems/symptoms:… " ; in the study, the investigators will ask : " Do you have any of the following stomach problems/symptoms : … ".
  With any of the 7 symptoms, the patient will be considered as symptomatic.
The proportions of patients answering "yes" to the clinical gastrointestinal symptoms questions were comparable at visit 3. | day 22
  The five-item PASS test is a valid tool for the evaluation of persistent acid-related symptoms in patients receiving PPI therapy. It demonstrates good content validity, test-retest reliability, responsiveness and construct validity in both English and French forms. The PASS test is a simple, clinically applicable tool for the identification of patients with persistent acid-related symptoms during therapy and the assessment of their responses to a change in therapy.
  The investigators will modifiy the first question for the study. While, it is usually asked: " Are you taking prescription medication for any of the following stomach problems/symptoms:… " ; in the study, the investigators will ask : " Do you have any of the following stomach problems/symptoms : … ".
  With any of the 7 symptoms, the patient will be considered as symptomatic.
The proportions of patients answering "yes" to the clinical gastrointestinal symptoms questions were comparable at visit 4. | day 29
  The five-item PASS test is a valid tool for the evaluation of persistent acid-related symptoms in patients receiving PPI therapy. It demonstrates good content validity, test-retest reliability, responsiveness and construct validity in both English and French forms. The PASS test is a simple, clinically applicable tool for the identification of patients with persistent acid-related symptoms during therapy and the assessment of their responses to a change in therapy.
  The investigators will modifiy the first question for the study. While, it is usually asked: " Are you taking prescription medication for any of the following stomach problems/symptoms:… " ; in the study, the investigators will ask : " Do you have any of the following stomach problems/symptoms : … ".
  With any of the 7 symptoms, the patient will be considered as symptomatic.

SECONDARY OUTCOMES:
The intensity of the acid rebound symptoms | day 8
  The entire modified-PASS test will be evaluated with respect to patients' responses to the individual question; For each symptom, its severity will be measured and scored (minimum score 0: patient has no symptoms; maximum score 4: patient has symptoms requiring supplemental medications and affecting sleep, eating, drinking and daily activities).
  The overall score will represent the consequence of the rebound acid symptoms.
The intensity of the acid rebound symptoms | day 15
  The entire modified-PASS test will be evaluated with respect to patients' responses to the individual question; For each symptom, its severity will be measured and scored (minimum score 0: patient has no symptoms; maximum score 4: patient has symptoms requiring supplemental medications and affecting sleep, eating, drinking and daily activities).
  The overall score will represent the consequence of the rebound acid symptoms.
The intensity of the acid rebound symptoms | day 22
  The entire modified-PASS test will be evaluated with respect to patients' responses to the individual question; For each symptom, its severity will be measured and scored (minimum score 0: patient has no symptoms; maximum score 4: patient has symptoms requiring supplemental medications and affecting sleep, eating, drinking and daily activities).
  The overall score will represent the consequence of the rebound acid symptoms.
The intensity of the acid rebound symptoms | day 29
  The entire modified-PASS test will be evaluated with respect to patients' responses to the individual question; For each symptom, its severity will be measured and scored (minimum score 0: patient has no symptoms; maximum score 4: patient has symptoms requiring supplemental medications and affecting sleep, eating, drinking and daily activities).
  The overall score will represent the consequence of the rebound acid symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Service de de médecine interne et de rehabilitation, Beau-séjour, HUG, Geneva
  - Service de réadaptation de l'appareil locomoteur Clinique romande de réadaptation, Sion, Sion

REFERENCES:
- [Result] Katz MH. Failing the acid test: benefits of proton pump inhibitors may not justify the risks for many users. Arch Intern Med. 2010 May 10;170(9):747-8. doi: 10.1001/archinternmed.2010.64. No abstract available. PMID 20458079
- [Result] Waldum HL, Arnestad JS, Brenna E, Eide I, Syversen U, Sandvik AK. Marked increase in gastric acid secretory capacity after omeprazole treatment. Gut. 1996 Nov;39(5):649-53. doi: 10.1136/gut.39.5.649. PMID 9026477
- [Result] Bjornsson E, Abrahamsson H, Simren M, Mattsson N, Jensen C, Agerforz P, Kilander A. Discontinuation of proton pump inhibitors in patients on long-term therapy: a double-blind, placebo-controlled trial. Aliment Pharmacol Ther. 2006 Sep 15;24(6):945-54. doi: 10.1111/j.1365-2036.2006.03084.x. PMID 16948806